CLINICAL TRIAL: NCT02192151
Title: The Pharmacokinetic and Bioavailability Studies of PHN131, an Oral Formulation of Nalbuphine Hydrochloride, in Healthy Volunteers
Brief Title: Study of PHN131 in Healthy Volunteers
Status: Terminated | Type: Observational
Why Stopped: CSR completed
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PH-CP019
Record Dates: First submitted 2013-11-24; First posted 2014-07-16 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Analgesia Disorder
Keywords: Analgesic; Narcotics; Opioids; Non-scheduled substanse

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the safety and to investigate the pharmacokinetic properties and bioavailability of PHN131 in healthy volunteers

DETAILED DESCRIPTION:
1. Efficacy endpoint(s): the pharmacokinetic properties and bioavailability of PHN131 The efficacy endpoint will be the pharmacokinetic properties after administered PHN131 such as the concentration of nalbuphine in plasma and pharmacokinetic parameters of PHN131 analyzed from the concentration of nalbuphine in plasma. The bioavailability of PHN131 will be calculated from the pharmacokinetic parameters of PHN131 and Nubain® injection.
2. Safety evaluation:

The safety evaluation will include the vital signs monitoring such as blood pressure, pulse rate, body temperature and respiratory rate in the treatment period.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in the study:

1. Normal healthy adult subjects between 20 to 40 years of age.
2. Body weight within 80 to 120% of ideal body weight. The ideal body weight is defined as: (subjects' height - 80) x 0.7
3. Acceptable medical history and physical examination including:

   * Normal chest X-ray and ECG results within six months prior to the Treatment Period of dose.
   * No particular clinical significance in general disease history within two months prior to the Treatment Period of dose.
4. Acceptable clinical laboratory determinations without significant deviation from normal values within two months prior to the Treatment Period of dose, which includes AST, ALT, garma-GT, alkaline phosphatase, total bilirubin, albumin glucose, BUN, uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology within two months prior to the study, which includes hemoglobin, hematocrit, red blood cells, MCV, MCH, MCHC, white blood cells and platelets.
6. Acepatable urinalysis within two months prior to the study, which includes pH, urine glucose and protein.
7. Signed the written informed consent to participate in this study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Recent history of drug or alcohol addiction or abuse.
2. A clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
3. History of allergic response(s) to nalbuphine or related drugs.
4. History of clinically significant allergies including drug allergies or allergic bronchial asthma.
5. Evidence of chronic or acute infectious disease.
6. Any clinically significant illness or surgery during the 4 weeks prior to the Treatment Period of dose (as determined by the clinical investigator).
7. Taking any drugs known to induce and/or inhibit hepatic drug metabolism within one month prior to the Treatment Period of dose.
8. Receiving any investigational drug within one month prior to the Treatment Period of dose.
9. Taking any prescription medication or any nonprescription medication within two weeks prior to the Treatment Period of dose.
10. Donating greater than 150 ml of blood within two months prior to the Treatment Period of dose or donating plasma (e.g. plasmapheresis) within 14 days prior to the Treatment Period of dose. All subjects will be advised not to donate blood for 4 weeks after completing the study.
11. Consumption of caffeine, xanthine-containing products (i.e. coffee, tea, caffeine-containing sodas, colas and chocolates, etc.) and/or alcohol at least 48 hours prior to day on which dosing is scheduled and during the periods when blood samples are being collected.
12. Any other medical reason(s) as determined by the clinical investigator.
13. Patient is pregnant or breastfeeding. Women of childbearing potential have positive urine pregnancy test at baseline.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint(s) | 10 days
  The pharmacokinetic properties and bioavailability of PHN131 The efficacy endpoint will be the pharmacokinetic properties after administered PHN131 such as the concentration of nalbuphine in plasma and pharmacokinetic parameters of PHN131 analyzed from the concentration of nalbuphine in plasma. The bioavailability of PHN131 will be calculated from the pharmacokinetic parameters of PHN131 and Nubain® injection.

SECONDARY OUTCOMES:
Safety evaluation | 10 days
  The safety evaluation will include the vital signs monitoring such as blood pressure, pulse rate, body temperature and respiratory rate in the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Shung-Tai Ho, Ph.D, Principal Investigator — Tri-service General Hospital & National Defense Medical Center
Locations (1):
- General Clinical Research Center, Tri-service General Hospital, Taipei, Taiwan